CLINICAL TRIAL: NCT04554888
Title: Characterization of New Human Models of Non-histaminergic Itch and Their Interaction With the TRPM8 Receptor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, PhD, Assistant Professor, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20200005 2nd project
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Itch
MeSH Terms: conditions — Pruritus | interventions — Doxepin; Papain; Histamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxepin Application (Experimental): During the session each forearm of the subject will be divided into four squared areas (2.5x2.5 cm), see Figure 4. Four of the areas will be treated with doxepin for 1 hour and 30 minutes (with a patch to deposit 1.2 grams of cream). Each patch will be covered with Tegaderm I.V., an occlusive, adhesive dressing (3M), for at least 1½ hours 48. At the end of the pre-treatment period, the patches will be removed and the skin will be cleaned with alcohol.
  Interventions: Drug: Doxepin Topical
- Itch Induction (Experimental): After Doxepin removal, Then tests with papain, cowhage, histamine or vehicle will be conducted. Each substance will be randomly applied in two areas, one pretreated with doxepin and one with no pre-treatment.
  Interventions: Drug: Papain; Drug: Histamine; Other: Cowhage

INTERVENTIONS:
Drug: Doxepin Topical — Four of the areas will be treated with doxepin for 1 hour and 30 minutes (with a patch to deposit 1.2 grams of cream). Each patch will be covered with Tegaderm I.V., an occlusive, adhesive dressing (3M), for at least 1½ hours
  Arms: Doxepin Application
Drug: Papain — Papain will be applied by 1 SPT prick thought the skin
  Arms: Itch Induction
Drug: Histamine — Histamine will be applied by 1 SPT prick thought the skin
  Arms: Itch Induction
Other: Cowhage — Cowhage spicules are 1-2 mm in length and have diameter of 1-3 µm at their tip. 30-35 spicules are gently rubbed into a 1 cm diameter skin area.
  Arms: Itch Induction

SUMMARY:
In this experiment the investigators would like to assess if papain induces an itch sensation comparable to the itch sensation induced by cowhage and to confirm that the mechanism of action of papain follows the non-histaminergic pathway.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other addictive drugs
* Previous or current history of neurological, dermatological, immunological musculoskeletal, cardiac disorder or mental illnesses that may affect the results (e.g. neuropathy, muscular pain in the upper extremities, etc.).
* Lack of ability to cooperate
* Current use of medications that may affect the trial such as antihistamines, antipsychotics and pain killers, as well as systemic or topical steroids.
* Skin diseases
* Moles, scars or tattoos in the area to be treated or tested.
* Hypersensitivity to papaya and mango fruit, cashew nuts, rubber latex
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Superficial blood perfusion | 15 minutes
  Superficial blood perfusion is measured by a Speckle contrast imager (FLPI, Moor Instruments, England).
Measuring itch intensity by computerized Visual Analog Scale Scoring | 15 minutes
  The subjects will rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable" and similarly for sensations of stinging/pricking and burning, both of which are frequently associated with the sensation of itch.
Measuring pain intensity by computerized Visual Analog Scale Scoring | 15 minutes
  The subjects will rate the sensation of pain on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no pain" and 100 indicates "worst pain imaginable".
Measuring Alloknesis | 15 minutes
  Alloknesis is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 milliNewton of force). This stimulator is applied 0.5 cm outside the area of itch provocation.

SECONDARY OUTCOMES:
Measurement of Cold Detection Thresholds (CDT) | 15 minutes
  The tests for thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature decreases 1°C per second from a starting temperature of 32°C until the subject perceives a temperature change (cold sensation) and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 0°C will be used.
Measurement of Cold PainThresholds (CPT) | 15 minutes
  The tests for thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature decreases 1°C per second from a starting temperature of 32°C until the subject perceives a temperature change (cold sensation) and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 0°C will be used.
Measurement of Heat Pain Thresholds (HPT) | 15 minutes
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature raises 1°C per second from a starting temperature of 32°C until the subject detects a painful sensation and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 52°C will be used.
Measurement of Warm Detection Thresholds (WDT) | 15 minutes
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature raises 1°C per second from a starting temperature of 32°C until the subject detects a painful sensation and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 52°C will be used.
Measurement of Pain to Supra-threshold Heat Stimuli | 15 minutes
  The tests will be conducted by using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. The subjects will have to rate the pain to two suprathreshold heat pain stimuli (starting and ending at 32°C with an increase and decrease of 5°C and 3 s plateau at 50°C).
Measurement of Mechanical Pain Thresholds (MPT) | 15 minutes
  This test is conducted using a pin-prick set (Aalborg University, Aalborg). This test is conducted using a pin-prick set (Aalborg University, Aalborg).easurement of Mechanical Pain Thresholds (MPT)
Measurement of Mechanical Pain Sensitivity (MPS) | 15 minutes
  This test is conducted using a pin-prick set (Aalborg University, Aalborg).
Touch Pleasantness (TP) | 15 minutes
  Pleasant touch sensation measured using astandardized sensory brush (SENSELab Brush-05, Somedic AB, Hörby, Sweden) exerting a force of 200 to 400 mN.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark